CLINICAL TRIAL: NCT03548597
Title: Evaluation of the Diagnostic of Hepatic Fibrosis With the XL Probe of the Fibroscan Versus Biopsies in Severe Obese Patients Candidates to Bariatric Surgery
Brief Title: Evaluation of the Diagnostic of Hepatic Fibrosis With the in Severe Obese Patients Candidates to Bariatric Surgery
Status: Completed | Type: Observational
Sponsor: European Georges Pompidou Hospital (Other)
Collaborators: Echosens (Industry)
Responsible Party: Principal Investigator, Charles Barsamian, Doctor of Medicine, European Georges Pompidou Hospital
Other Study IDs: B047
Record Dates: First submitted 2018-05-24; First posted 2018-06-07 (Actual); Last update posted 2018-06-07 (Actual); Status verified 2018-06

CONDITIONS: Steatosis; Obesity; Fibrosis, Liver
MeSH Terms: conditions — Fatty Liver; Obesity; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Evaluation of the Diagnostic of Hepatic Fibrosis With the XL Probe of the Fibroscan Versus Biopsies in Severe Obese Patients Candidates to Bariatric Surgery — Evaluation of the Diagnostic of Hepatic Fibrosis With the XL Probe of the Fibroscan Versus Biopsies in Severe Obese Patients Candidates to Bariatric Surgery

SUMMARY:
Background:

The XL probe of FibroScan was recently developed to realize liver stiffness measurements (LSM) in overweight patients.

Severe obese patients have a high prevalence of liver injuries and could benefit of liver evaluation prior to bariatric surgery.

Objectives:

Assess the FibroScan applicability, reliability and diagnostic performances in severe obese patients' candidates for bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* Severe obese patients candidate to bariatric surgery with no history of liver disease have a large prevalence of liver lesions.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Severe obese patients candidate to bariatric surgery
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2012-04-04 (Actual); Primary Completion 2015-01-12 (Actual); Study Completion 2016-12-06 (Actual)

PRIMARY OUTCOMES:
Elasticity measured with the Fibroscan XL | 3 years
  Liver elasticity will be measured non-invasively with Fibroscan. As this is a non-invasive measure, no adverse effects are expected. No treatment planned.

SECONDARY OUTCOMES:
53/5000 Evolution of elasticity after bariatric surgery | 3 years
  The evolution of elasticity will be measured non-invasively with fibroscan after bariatric surgery. NO adverse effects are expected in relation to this measure.

REFERENCES:
- [Derived] Barsamian C, Carette C, Sasso M, Poghosyan T, Bedossa P, Emile JF, Parlier D, Miette V, Bouillot JL, Czernichow S, Rives-Lange C. Diagnostic of hepatic fibrosis with the XL probe of the Fibroscan versus biopsies in patients candidates to bariatric surgery. Clin Nutr ESPEN. 2020 Jun;37:226-232. doi: 10.1016/j.clnesp.2020.02.010. Epub 2020 Mar 12. PMID 32359748